CLINICAL TRIAL: NCT00987194
Title: HIV Testing in the Emergency Department at Baystate Medical Center: A Pilot Program Version 1.5, May 2009
Brief Title: HIV Testing in the Emergency Department at Baystate Medical Center: A Pilot Program
Status: Completed | Type: Observational
Sponsor: Baystate Medical Center (Other)
Collaborators: Massachusetts Department of Health (Other Government)
Responsible Party: Daniel Skiest, MD, Baystate Medical Center
Other Study IDs: IRB09-012
Record Dates: First submitted 2009-09-25; First posted 2009-09-30 (Estimated); Last update posted 2010-07-14 (Estimated); Status verified 2010-07

CONDITIONS: HIV Infections
Keywords: HIV; rapid testing; HIV seronegativity
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Background Recently, the CDC issued recommendations calling for HIV screening for patients aged 13-64, when the individual accesses the health care system. For many patients, the emergency department (ED) is the primary or only contact point for health care. The rapid HIV test can be done as a point of care test in the ED.

Study Objectives

A. Primary:

1. To initiate HIV testing in the Baystate ED.

B. Secondary:

1. To estimate the resources involved in initiating a rapid HIV testing program in the ED.
2. To describe the process of initiating a rapid HIV testing program.
3. To compare the yield of testing for HIV in patients with known HIV risk factors compared to those without known risk factors.
4. To describe the characteristics of the population tested for HIV in the ED.
5. To determine the number of patients who declined testing and the reasons for declining testing.
6. To analyze ED staff attitudes re: HIV rapid testing in the ED.

Methods A trained HIV Educator/counselor will approach patients in the ED to offer free rapid HIV testing, at a time they are not currently engaged with the health care provider. Study informed consent and HIV consent will be obtained prior to testing. The HIV educator will obtain demographic and clinical information on the enrolled subjects including prior HIV testing and HIV risk factors. Patients testing negative will be counseled regarding HIV risk reduction strategies. Patients with an initial positive rapid HIV test will have blood drawn for confirmation (Western Blot) and will be referred to an HIV clinic for follow-up and treatment. Additionally, to assess acceptability of rapid testing in the ED, a brief anonymous electronic survey will be conducted of health care providers in the ED prior to starting this pilot program and following the program.

Data Analysis The yield of testing will be calculated as will the seroprevalence of those tested. Among patients who decline HIV testing but agree to study participation (sign consent form), the number refusing testing will be recorded and reasons for refusing will be analyzed. The yield of testing will be compared in patients with to those without known HIV risk factors.

DETAILED DESCRIPTION:
I. Background Recently, CDC issued recommendations calling for HIV screening for patients aged 13-64, when the individual accesses the health care system 1. For many patients, especially those without a primary care provider, the emergency department (ED) is the primary or only contact point for the health care system. Testing individuals while they are in the ED has the potential to identify persons who do not perceive themselves to be at risk for HIV. Several academic EDs have begun to offer HIV testing 10, and have initially indicated promising results.

II. Rationale for testing in ED Testing in the ED has several potential advantages. It leads to shorter hospital stays, increases the number of newly diagnosed patients with HIV who are discharged from the hospital aware of their HIV status, and improved entry into outpatient care for patients admitted at the time of their initial HIV diagnosis. Another advantage of HIV testing in the ED is the ability to link newly diagnosed patients to an HIV clinician.

The optimal approach to testing for HIV in the ED is not known. Testing without risk assessment can identify persons with undiagnosed HIV infection and reduce reluctance assessing risk behavior.

While widespread routine HIV screening (e.g. testing as many patients as possible presenting to the ED) is likely to result in the highest number of positive tests, this strategy is expensive, burdensome and will not be practical in a busy city ED. In the setting of limited resources, a strategy of targeted testing (testing patients with established risk factors for HIV) may be a more cost-effective strategy. It may also be more practical and may be more acceptable to ED staff.

Another issue which needs further study is identifying the optimal personnel to conduct rapid HIV testing in the ED. There are advantages and disadvantages to requiring ED staff to counsel and consent patients for HIV testing. The ED staff may believe the testing is not in their purview and may not believe they have time to devote to testing.

Another important issue is the feasibility of conducting rapid testing in the ED. How many individuals can be tested in an eight hour day by one HIV educator? What are the barriers to conducting rapid testing in the ED and what solutions can be implemented to overcome these barriers? Finally, what are the attitudes of the ED staff regarding HIV testing in the ED? By collecting data during the implementation of this pilot project we hope to optimize the approach to HIV testing in the ED.

III. Hypothesis

Primary - Initiation of a rapid HIV testing program in the ED of a community teaching hospital is feasible but will require substantial resources and cooperation between multiple departments and stakeholders.

Secondary- Patients with known HIV risk factors will have a higher HIV seroprevalence compared to patients without known risk factors.

IV. Study Objectives

A. Primary:

1. To initiate HIV testing in the Baystate ED in order to increase the number of new HIV diagnoses and to link these patients to HIV care.

B. Secondary:

1. To estimate the resources involved in initiating a rapid HIV testing program in the ED of a large community teaching hospital.
2. To describe the process of initiating a rapid HIV testing program and the barriers to implementation.
3. To compare the yield of HIV testing in patients with known HIV risk factors compared to those without known risk factors in patients presenting to the ED in order to estimate the feasibility of a random screening strategy compared to a targeted screening strategy.
4. To describe the characteristics of the population tested for HIV in the ED.
5. To determine the number of patients who decline testing and the reasons for declining testing.

   .
6. To determine the number of newly diagnosed individuals who were successfully linked to an HIV provider and the number who received antiretroviral therapy within one year of initial diagnosis.
7. To analyze ED staff attitudes re: HIV rapid testing in the ED

V. Methods:

Overview of Operations:

A trained HIV Health Educator will offer HIV counseling and testing to ED patients interested in HIV testing. The number of patients studied will be determined by how many patients can be approached by the HIV Health Educator.

Following initial counseling the HIV Health educator will obtain an Informed Consent for study participation and HIV testing as well as HIPPA authorization from the study participants. Patients who decline testing will be asked to consent to participate in the study by signing a research consent form and will be asked the reason(s) they decline testing. The reasons for declining testing will be recorded among those who agree to participate.

ED patients may also be referred to the HIV Health Educator by the ED nurse or clinician (physician or midlevel clinician) if the nurse or clinician believes HIV testing is indicated based on potential risk factors for HIV or conditions possibly related to (as a part of the patient's social and medical history). Finally, a patient who is an ED patient (and has not otherwise been approached for testing) may also request to be tested for HIV while in the ED.

After identification of potential patients according to one of the above methods, the health educator will approach patients who are not otherwise engaged with an ED staff person and prior to discharge from the ED. Patients will be approached in a fashion that does not interfere with the normal flow of the ED visit. Patients too ill to approach (in the opinion of the HIV health educator or ED staff) will be excluded, as will patients who have previously tested positive for HIV. The HIV Health Educator will do an initial risk assessment and brief pretest counseling prior to obtaining verbal and written consent for HIV testing. Counseling and consent will be in Spanish for patients whose primary language is Spanish. (A consent form will be translated into Spanish.) The Health Educator will then obtain blood via finger stick from the patient. The test will be run (according to the instructions in the package insert) by the Health Educator in a designated area of the ED. Results will be read as reactive or non-reactive. In the event of a non-reactive test the patient will be informed of the result. During the post-test counseling session patients will be given risk reduction information and shown harm reduction skills and techniques and counseled on appropriate behaviors to minimize risk of HIV acquisition. The patient will also be offered an opportunity to be retested in the future and encouraged to visit an I-CTR program for sexually transmitted disease and hepatitis testing and vaccinations as needed. Testing will be entirely voluntary and will be confidential

In case of a reactive rapid test the client will be brought to the consultation room in the ED to ensure privacy and will be informed that the result is a preliminary reactive result for HIV and that a confirmatory test is required. In the case of a reactive test (initial positive), a venous blood sample will be drawn by the HIV Health Educator for confirmation via HIV Western blot. The HIV Health Educator is licensed to draw blood. A separate written consent for HIV will be obtained prior to obtaining blood for the HIV Western blot. The Western blot will be sent to the MA State laboratory with an expected result in < 5 business days. The results of the initial test and the confirmatory test will not be entered into the patient medical record. The state of Massachusetts Department of Health will not have the names of patients tested. The only reporting to the state of positive HIV results will be done when the patient accesses medical care as per state law e.g. the patient's health care provider will report the results to the state. This reporting is not part of this study.

The HIV health educator has extensive experience in informing patients/clients of positive HIV test results and has a plan in place to counsel such patients. The PI or his representative will also be available to counsel patients with a positive HIV test result. In the rare case of a catastrophic emotional reaction to a positive test result the HIV health educator will involve the crisis team (Behavioral Health Network (BHN) Crisis Services). The BHN crisis services team is stationed in the ED and has experience counseling patients who are severely emotionally distraught. The BHN crisis team is aware of the HIV rapid testing program and is willing to participate when needed. If the patient has problems after he/she leaves the ED, he/she will be able to contact the HIV health educator who, in conjunction with the PI, can then make a referral (if needed) for psychological/psychiatric follow-up. Once the patient has followed up with a health care provider in the HIV/ID clinic (generally within 5 days) (see below for details) if psychological issues arise that health care provider will make an appropriate referral to a mental health provider.

In cases where the rapid HIV test is reactive, the HIV Health Educator will be responsible for linking the patient to appropriate medical care. An appointment in the HIV/ID clinic will be given to the patient prior to discharge from the ED.

The patient can be referred to any of the three Baystate Health Centers In the event where the tested patient leaves the ED prior to receipt of test results the counselor will notify the patient by phone or mail to schedule an appointment for receipt of results. A supportive referral for mental health assessment and counseling will also be made, as needed (see above).

Survey Prior to the start of rapid HIV testing in the ED, a brief electronic survey (using Survey Monkey software) will be conducted. The survey will be sent via email to ED physicians and midlevel providers. The survey instructions will explain that the survey is voluntary and confidential and that participants will not be identified. The same survey will be sent to the same individuals after the first six months of this pilot program to assess any changes in attitudes.

VI. Data Management/Security

The HIV Health Educator will collect data for clinical and study purposes. Data will be stored in paper records, not electronically. All patient information will be kept in individual folders by barcode. A barcode is assigned to each patient and is used as a specific identifier for each specimen tested. Once testing had been completed these folders will be stored in a locked file in the office of the principal investigator. There is a policy in place to maintain confidentiality and privacy throughout the entire testing process: written consent, test performance, disclosure of test results, and storage of records. We will not allow access to other researchers or answer any other questions without IRB approval. All files will be kept for seven years.

VII. ANALYSIS PLAN

Demographic information obtained from the patient at the time of testing as part of the pilot testing will be recorded on a data collection sheet. Data collected will include risk factors for HIV, ethnicity, sex, age, payer status, zip code, homeless status, prior testing status (and dates of prior testing), co-morbid medical conditions possibly related to HIV diagnosis and chief complaint on presentation to ED. In addition, general demographic information about patients admitted to the ED during the study period will be requested and de-identified and, if appropriate, will be extrapolated for calculation of seroprevalence e.g. the characteristics of the patients tested for HIV will be compared to the overall ED population in order to ascertain whether the tested sample is representative of the ED population.

The number of patients approached for testing will be recorded as will the total number of patients registered in the ED during the period of testing (eight hours per day, five days per week). The number of reactive tests as well as the number of positive confirmatory tests will be determined. In order to determine the yield of testing and to estimate seroprevalence in the ED, the number of patients testing positive (confirmed by Western blot) will be divided by the total number tested. Further calculations will incorporate the yield of testing in those with risk factors and compare to those with no reported risk factors. In addition, the number of patients with reactive tests attending an initial and subsequent HIV clinic visit as well as the number presenting with an AIDS diagnosis and the number commencing antiretroviral therapy within one year after testing will be recorded.

The HIV health educator will observe and record barriers to testing in the ED staff.. Modifications in the testing policy will be implemented based on the assessment of the HIV health educator in order to maximize the number of patients tested. No identifying information concerning ED staff members will be recorded. Modifications in the testing policy will be implemented based on this assessment in order to maximize the number of patients tested.

In order to ascertain the sustainability of the program, following the initial pilot program, the cost of HIV testing will be estimated by including the following costs: health educator salary plus benefits, program administration, materials, test kits, postage and confirmatory testing. The cost per test, cost per approached patient, cost per enrolled patient, and cost per confirmed infection detected will be calculated, as will the annualized direct cost.

Results of the survey will be tallied. Pre and post surveys will be compared using Chi square for categorical data (e.g. for yes, no questions) and Student's T test for continuous data.

Data from the main study will be entered into Microsoft Excel. StatView statistical software will be used to analyze data. Categorical data will be analyzed by the appropriate test e.g. Chi Square or Fisher's exact test. Continuous data will be analyzed using the Student's T-test.

ELIGIBILITY:
Inclusion Criteria:

* Emergency department patients aged 18 years or older, appropriate for HIV testing will be identified by the HIV health educator.
* Patients who are not otherwise occupied and who are not known to be HIV+ will be approached for consent to the study and for rapid HIV testing.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Emergency department patients aged 18 years or older
Sampling Method: Non-Probability Sample
Enrollment: 1087 (Actual)
Dates: Start 2009-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
The feasibility of initiating a rapid HIV testing program in the emergency department of a community teaching hospital in an a medium size city. | 2 years

SECONDARY OUTCOMES:
To determine the number of newly diagnosed individuals who were successfully linked to an HIV provider and the number who received antiretroviral therapy within one year of initial diagnosis. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Skiest, MD, Principal Investigator — Baystate Medical Center
Locations (1):
- Baystate Medical Center, Springfield, Massachusetts, United States

REFERENCES:
- [Background] Branson BM, Handsfield HH, Lampe MA, Janssen RS, Taylor AW, Lyss SB, Clark JE; Centers for Disease Control and Prevention (CDC). Revised recommendations for HIV testing of adults, adolescents, and pregnant women in health-care settings. MMWR Recomm Rep. 2006 Sep 22;55(RR-14):1-17; quiz CE1-4. PMID 16988643
- [Background] Palella FJ Jr, Deloria-Knoll M, Chmiel JS, Moorman AC, Wood KC, Greenberg AE, Holmberg SD; HIV Outpatient Study Investigators. Survival benefit of initiating antiretroviral therapy in HIV-infected persons in different CD4+ cell strata. Ann Intern Med. 2003 Apr 15;138(8):620-6. doi: 10.7326/0003-4819-138-8-200304150-00007. PMID 12693883
- [Background] Keiser P, Nassar N, Kvanli MB, Turner D, Smith JW, Skiest D. Long-term impact of highly active antiretroviral therapy on HIV-related health care costs. J Acquir Immune Defic Syndr. 2001 May 1;27(1):14-9. doi: 10.1097/00126334-200105010-00003. PMID 11404515
- [Background] Centers for Disease Control and Prevention (CDC). False-positive oral fluid rapid HIV tests--New York City, 2005-2008. MMWR Morb Mortal Wkly Rep. 2008 Jun 20;57(24):660-5. PMID 18566566
- [Background] Hutchinson AB, Branson BM, Kim A, Farnham PG. A meta-analysis of the effectiveness of alternative HIV counseling and testing methods to increase knowledge of HIV status. AIDS. 2006 Aug 1;20(12):1597-604. doi: 10.1097/01.aids.0000238405.93249.16. PMID 16868440
- [Background] Lubelchek R, Kroc K, Hota B, Sharief R, Muppudi U, Pulvirenti J, Weinstein RA. The role of rapid vs conventional human immunodeficiency virus testing for inpatients: effects on quality of care. Arch Intern Med. 2005 Sep 26;165(17):1956-60. doi: 10.1001/archinte.165.17.1956. PMID 16186464
- [Background] Marks G, Crepaz N, Senterfitt JW, Janssen RS. Meta-analysis of high-risk sexual behavior in persons aware and unaware they are infected with HIV in the United States: implications for HIV prevention programs. J Acquir Immune Defic Syndr. 2005 Aug 1;39(4):446-53. doi: 10.1097/01.qai.0000151079.33935.79. PMID 16010168
- [Background] Holtgrave DR. Costs and consequences of the US Centers for Disease Control and Prevention's recommendations for opt-out HIV testing. PLoS Med. 2007 Jun;4(6):e194. doi: 10.1371/journal.pmed.0040194. PMID 17564488
- [Background] Bogart LM, Howerton D, Lange J, Setodji CM, Becker K, Klein DJ, Asch SM. Provider-related barriers to rapid HIV testing in U.S. urban non-profit community clinics, community-based organizations (CBOs) and hospitals. AIDS Behav. 2010 Jun;14(3):697-707. doi: 10.1007/s10461-008-9456-3. Epub 2008 Sep 3. PMID 18770022
- [Background] Ehrenkranz PD, Ahn CJ, Metlay JP, Camargo CA Jr, Holmes WC, Rothman R. Availability of rapid human immunodeficiency virus testing in academic emergency departments. Acad Emerg Med. 2008 Feb;15(2):144-50. doi: 10.1111/j.1553-2712.2008.00028.x. PMID 18275444
- [Background] Centers for Disease Control and Prevention (CDC). Missed opportunities for earlier diagnosis of HIV infection--South Carolina, 1997-2005. MMWR Morb Mortal Wkly Rep. 2006 Dec 1;55(47):1269-72. PMID 17136020
- [Background] Rothman RE, Ketlogetswe KS, Dolan T, Wyer PC, Kelen GD. Preventive care in the emergency department: should emergency departments conduct routine HIV screening? a systematic review. Acad Emerg Med. 2003 Mar;10(3):278-85. doi: 10.1111/j.1553-2712.2003.tb02004.x. PMID 12615596